CLINICAL TRIAL: NCT04433442
Title: Post-Marketing Surveillance to Evaluate the Safety and Effectiveness of Risankizumab (Skyrizi) in Adult Moderate to Severe Plaque Psoriasis and Psoriatic Arthritis Patients
Brief Title: Study to Assess the Safety and Change in Disease Symptoms of Risankizumab (Skyrizi) in Adult Participants With Moderate to Severe Plaque Psoriasis and Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-271
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: Psoriasis; Plaque Psoriasis; Psoriatic Arthritis; Risankizumab; Skyrizi; Prefilled syringe
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Moderate to Severe Plaque Psoriasis or Psoriatic Arthritis: Participants will receive risankizumab as prescribed by the physician in routine clinical practice.

SUMMARY:
Plaque Psoriasis is a chronic inflammatory disease in which skin cells build up and develop scaly red and white patches on the skin. Psoriatic arthritis (PsA) is a type of arthritis (swelling and stiffness in the joints) that is frequently seen in trial participants who also have the skin condition psoriasis. It is caused by an overactive immune system where the body attacks healthy tissue by mistake. This study will evaluate how safe risankizumab is for the treatment of plaque psoriasis or psoriatic arthritis and to assess change in disease symptoms.

Risankizumab is an approved drug for the treatment of psoriasis and psoriatic arthritis. Around 3000 adult participants with a moderate to severe plaque psoriasis or psoriatic arthritis who had been prescribed risankizumab by their doctor will be enrolled in this study in multiple sites across Korea. The sample size for this study is a requirement by local authorities.

Participants will receive risankizumab prefilled syringe for injection for 52 weeks as prescribed by their physician.

There is expected to be no additional burden for participants in this study. All study visits will occur during routine clinical practice and participants will be followed for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for the treatment with risankizumab according to the approved local label.
* Voluntarily agree to participate in this study and sign informed consent.

Exclusion Criteria:

- Contraindications to risankizumab as listed on the approved local label.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderate to severe plaque psoriasis or psoriatic arthritis
Sampling Method: Probability Sample
Enrollment: 2324 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Reported Adverse Events | Up to Week 72
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (63):
- South Korea (63):
  - Inje University - Busan Paik Hospital /ID# 238911, Busan, Busan Gwang Yeogsi
  - Inje University Haeundae Hospital /ID# 238933, Busan, Busan Gwang Yeogsi
  - Pusan National University Hospital /ID# 238896, Busan, Busan Gwang Yeogsi
  - Dankook University Hospital /ID# 223995, Cheonan-si, Chungcheongnam-do
  - SoonChunHyang University Hospital Cheonan /ID# 238909, Cheonan-si, Chungcheongnam-do
  - Kyungpook National University Hospital /ID# 238915, Daegu, Daegu Gwang Yeogsi
  - Chungnam National University Hospital /ID# 223993, Daejeon, Daejeon Gwang Yeogsi
  - Konyang University Hospital /ID# 238899, Daejeon, Daejeon Gwang Yeogsi
  - Kangwon National University Hospital /ID# 238902, Chuncheon, Gang Weondo
  - Korea University Ansan Hospital /ID# 223989, Ansan-si, Gyeonggido
  - Soon Chun Hyang University Hospital Bucheon /ID# 238894, Bucheon-si, Gyeonggido
  - The Catholic University Of Korea, Bucheon St. Mary'S Hospital /ID# 270826, Bucheon-si, Gyeonggido
  - Hallym University Dongtan Sacred Heart Hospital /ID# 238927, Hwaseong, Gyeonggido
  - Dongguk University Ilsan Hospital /ID# 259337, Ilsan, Gyeonggido
  - Gachon University Gil Medical Center /ID# 262788, Incheon, Gyeonggido
  - Catholic Kwandong University International St.Mary's Hospital /ID# 262855, Incheon, Gyeonggido
  - CHA Bundang Medical Center /ID# 238916, Seongnam, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 238900, Seongnam-si, Gyeonggido
  - Hallym University Sacred Heart Hospital /ID# 238913, Seoul, Gyeonggido
  - Hallym University Sacred Heart Hospital /ID# 238930, Seoul, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 248371, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 238920, Suwon, Gyeonggido
  - Uijeongbu Eulji Medical Center - Eulji University /ID# 259200, Uijeongbu-si, Gyeonggido
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital /ID# 259201, Uijeongbu-si, Gyeonggido
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital /ID# 259202, Uijeongbu-si, Gyeonggido
  - Yongin Severance Hospital /ID# 238925, Yŏngin, Gyeonggido
  - Daegu Catholic University Medical Center /ID# 238921, Daegu, Gyeongsangbuk-do
  - Keimyung University Dongsan Hospital /ID# 238932, Daegu, Gyeongsangbuk-do
  - Dongguk University Gyeongju Hospital /ID# 238923, Gyeongju, Gyeongsangbuk-do
  - Pusan National University Yangsan Hospital /ID# 259098, Yangsan, Gyeongsangnam-do
  - The Catholic University of Korea, Incheon St. Mary's Hospital /ID# 238934, Incheon, Incheon Gwang Yeogsi
  - Inha University Hospital /ID# 248373, Incheon, Incheon Gwang Yeogsi
  - Wonkwang University Hospital /ID# 238901, Iksan, Jeonrabugdo
  - Design Hospital /ID# 238929, Jeollabuk-do, Jeonrabugdo
  - Chosun University Hospital /ID# 238910, Gwangju, Jeonranamdo
  - Chonnam National University Hospital /ID# 259199, Gwangju, Jeonranamdo
  - Chungbuk National University Hospital /ID# 238891, Cheongju-si, North Chungcheong
  - Chungang University Hospital /ID# 238918, Dongjak-gu, Seoul Teugbyeolsi
  - Inje University Sanggye Paik Hospital /ID# 238903, Seoul, Seoul Teugbyeolsi
  - Nowon Eulji Medical Center, Eulji University /ID# 259198, Seoul, Seoul Teugbyeolsi
  - Seoul Medical Center /ID# 238906, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Hospital /ID# 248375, Seoul, Seoul Teugbyeolsi
  - Korea University Anam Hospital /ID# 238931, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 238904, Seoul, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 238908, Seoul, Seoul Teugbyeolsi
  - National Medical Center /ID# 238917, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center /ID# 223996, Seoul, Seoul Teugbyeolsi
  - VHS(Veterans Health Service) Medical Center /ID# 238935, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 238912, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital /ID# 223990, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 238919, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 248370, Seoul, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 238922, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Yeouido ST. Mary's Hospital /ID# 248372, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 262789, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 270776, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital /ID# 238905, Seoul, Seoul Teugbyeolsi
  - Kyungpook National University Chilgok Hospital /ID# 238914, Daegu
  - Yeungnam University Medical Center /ID# 238924, Daegu
  - Yonsei University Health System Severance Hospital /ID# 238928, Seoul
  - Duplicate_Kyunghee University Hospital at Gangdong /ID# 248369, Seoul
  - Hallym University Kangdong Sacred Heart Hospital /ID# 238936, Seoul
  - Hallym University Kangdong Sacred Heart Hospital /ID# 238937, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/